CLINICAL TRIAL: NCT00931580
Title: Supplemental Vitamin D and Functional Outcomes in Early Adolescence
Brief Title: Vitamin D Needs of Early Adolescent Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: Purdue University (Other); Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Dr. Richard D. Lewis, Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 1R01HD57126-01A2 UGA; 1R01HD057126-01A2 (NIH)
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Vitamin D; Adolescent; African American; White
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): placebo tablet
  Interventions: Dietary Supplement: Vitamin D3
- 400 IU (Experimental): Vitamin D3 tablet, 400 IU
  Interventions: Dietary Supplement: Vitamin D3
- 1,000 IU (Experimental): Vitamin D3 tablet, 1,000 IU
  Interventions: Dietary Supplement: Vitamin D3
- 2,000 IU (Experimental): Vitamin D3 tablet, 2,000 IU
  Interventions: Dietary Supplement: Vitamin D3
- 4,000 IU (Experimental): Vitamin D3 tablet, 4,000 IU
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — vitamin D3 supplementation at 400 IU vs 1,000 IU vs 2,000 IU vs 4,000 IU vs placebo for 12-weeks

SUMMARY:
While a large percentage of children have low blood vitamin D levels, the significance of these low levels and the impact on health is unclear. The purpose of this project is to determine the effects of varying doses of vitamin D supplementation over 12 weeks on blood indicators of health in white and black children, aged 9 to 13 years, from both the northern and southern US.

DETAILED DESCRIPTION:
Vitamin D intakes in children do not meet current US Dietary Reference Intake recommendations and emerging evidence suggests that a significant number of children, particularly those with darker skin pigmentation, have inadequate levels of serum 25-hydroxyvitamin D [25(OH)D]. The optimum level of circulating 25(OH)D has not been clearly defined in children, nor is it known what functional outcome measures are ideal for defining this level, or if these requirements would differ by race. Graded doses of vitamin D3 supplementation will be used in this dual-site, 12-week trial. The investigators hypothesize that a dose-response relationship will be observed between vitamin D supplementation and intermediate endpoints of skeletal health, and that race will modify these responses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-Hispanic
* Male, 10-13 years of age or female 9-11 years of age
* Within genitalia or breast stage 2/3
* Willing to provide blood/urine samples
* Free from taking vitamin, mineral or herbal supplements
* Able to swallow tablets

Exclusion Criteria:

* Menarche (females)
* Known bone diseases or disease known to influence bone metabolism (e.g. cerebral palsy, intestinal malabsorption, juvenile rheumatoid arthritis)
* Known growth disorder
* The use of medications that influence bone metabolism (e.g. corticosteroids, Attention Deficit Hyperactivity Disorder (ADHD) medications).

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 323 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
serum 25(OH)D | 0 weeks
PTH | 0 weeks
1,25(OH)2D | 0 weeks
fractional calcium absorption | 0 weeks
biochemical markers of bone turnover | 0 weeks
serum 25(OH)D | 3 weeks
serum 25(OH)D | 6 weeks
serum 25(OH)D | 9 weeks
serum 25(OH)D | 12 weeks
PTH | 3 weeks
PTH | 6 weeks
PTH | 9 weeks
PTH | 12 weeks
1,25(OH)2D | 3 weeks
1,25(OH)2D | 6 weeks
1,25(OH)2D | 9 weeks
1,25(OH)2D | 12 weeks
fractional calcium absorption | 12 weeks
biochemical markers of bone turnover | 3 weeks
biochemical markers of bone turnover | 6 weeks
biochemical markers of bone turnover | 9 weeks
biochemical markers of bone turnover | 12 weeks

SECONDARY OUTCOMES:
sunlight exposure | 0 weeks
dietary data | 0 weeks
physical activity data | 0 weeks
serum and urinary calcium | 0 weeks
body composition | 0 weeks
sunlight exposure | 3 weeks
sunlight exposure | 6 weeks
sunlight exposure | 9 weeks
sunlight exposure | 12 weeks
dietary data | 3 weeks
dietary data | 6 weeks
dietary data | 9 weeks
dietary data | 12 weeks
physical activity data | 3 weeks
physical activity data | 6 weeks
physical activity data | 9 weeks
physical activity data | 12 weeks
serum and urinary calcium | 3 weeks
serum and urinary calcium | 6 weeks
serum and urinary calcium | 9 weeks
serum and urinary calcium | 12 weeks
body composition | 3 weeks
body composition | 6 weeks
body composition | 9 weeks
body composition | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Lewis, PhD, Principal Investigator — The University of Georgia
Locations (3):
- United States (3):
  - The University of Georgia Dept of Foods & Nutrition, Athens, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Purdue University, West Lafayette, Indiana

REFERENCES:
- [Result] Lewis RD, Laing EM, Hill Gallant KM, Hall DB, McCabe GP, Hausman DB, Martin BR, Warden SJ, Peacock M, Weaver CM. A randomized trial of vitamin D(3) supplementation in children: dose-response effects on vitamin D metabolites and calcium absorption. J Clin Endocrinol Metab. 2013 Dec;98(12):4816-25. doi: 10.1210/jc.2013-2728. Epub 2013 Oct 3. PMID 24092833
- [Derived] Wright CS, Laing EM, Pollock NK, Hausman DB, Weaver CM, Martin BR, McCabe GP, Peacock M, Warden SJ, Hill Gallant KM, Lewis RD. Serum 25-Hydroxyvitamin D and Intact Parathyroid Hormone Influence Muscle Outcomes in Children and Adolescents. J Bone Miner Res. 2018 Nov;33(11):1940-1947. doi: 10.1002/jbmr.3550. Epub 2018 Aug 27. PMID 30001469
- [Derived] Giudici KV, Kindler JM, Martin BR, Laing EM, McCabe GP, McCabe LD, Hausman DB, Martini LA, Lewis RD, Weaver CM, Peacock M, Hill Gallant KM. Associations among osteocalcin, leptin and metabolic health in children ages 9-13 years in the United States. Nutr Metab (Lond). 2017 Mar 7;14:25. doi: 10.1186/s12986-017-0171-9. eCollection 2017. PMID 28286536
- [Derived] Ferira AJ, Laing EM, Hausman DB, Hall DB, McCabe GP, Martin BR, Hill Gallant KM, Warden SJ, Weaver CM, Peacock M, Lewis RD. Vitamin D Supplementation Does Not Impact Insulin Resistance in Black and White Children. J Clin Endocrinol Metab. 2016 Apr;101(4):1710-8. doi: 10.1210/jc.2015-3687. Epub 2016 Feb 17. PMID 26885880
- [Derived] Hill KM, Laing EM, Hausman DB, Acton A, Martin BR, McCabe GP, Weaver CM, Lewis RD, Peacock M. Bone turnover is not influenced by serum 25-hydroxyvitamin D in pubertal healthy black and white children. Bone. 2012 Oct;51(4):795-9. doi: 10.1016/j.bone.2012.06.014. Epub 2012 Jun 28. PMID 22750015